CLINICAL TRIAL: NCT00312949
Title: Consumer Internet Education About Mental Health Quality
Brief Title: Effectiveness of an Interactive Educational Website for Improving the Quality of Mental Health Care for People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald Steinwachs, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01MH067189 (NIH); R01MH067189 (NIH); DSIR 82-SEDR
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Patient participation; Patient education; Consumer involvement
MeSH Terms: conditions — Schizophrenia; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will use the interactive website
  Interventions: Behavioral: Interactive Website on management of schizophrenia
- 2 (Active Comparator): Participants will read written materials and watch a video
  Interventions: Behavioral: Written materials and video on management of schizophrenia

INTERVENTIONS:
Behavioral: Interactive Website on management of schizophrenia — Participants in the web-user group will sit with a laptop computer, answer questions about themselves and their treatment, receive feedback on care that may be inconsistent with current recommendations, and receive suggestions on how to discuss this with their physicians.
  Arms: 1
Behavioral: Written materials and video on management of schizophrenia — Participants in the written materials/video group will be given the reading material and will watch a 20-minute video.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of an interactive educational website in enhancing discussions about treatment issues and improving the quality of care for people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a disabling mental disorder that causes hallucinations and delusions in those affected by it. Research has proven that certain treatment methods are more effective in treating schizophrenia than others. However, not everyone with schizophrenia responds to treatment in the same way, and not all physicians use the same treatment methods. Educating individuals with schizophrenia about all treatments available instead of only the treatments they are receiving may improve the quality of care and lead to better correlation between treatment and quality standards. This study will evaluate the effectiveness of an interactive educational website in enhancing discussions about treatment issues and improving the congruence between expected quality of treatment and treatment received among people with schizophrenia.

Participants in this open label study will be randomly assigned to either use the interactive website or read written materials and watch a video. All three sources will contain information about evidence-based treatment recommendations. Both groups will complete a brief interview before performing their assigned tasks. Upon completion of the interview, participants in the written materials/video group will be given the reading material and will watch a 20-minute video. Participants in the web-user group will sit with a laptop computer, answer questions about themselves and their treatment, receive feedback on care that may be inconsistent with current recommendations, and receive suggestions on how to discuss this with their physicians. Participants in clinical settings will be asked to allow their next clinician visit to be audiotaped to assess outcomes. A phone interview will be conducted with all participants 2 months following the intervention to assess treatment satisfaction and other outcomes. Medical records will be reviewed to collect treatment information 6 months before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Able to read and write English
* Scheduled to see a participating clinician at one of the study sites

Exclusion Criteria:

* N/A

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Concordance of treatment with evidence-based recommendations | Measured at Month 6

SECONDARY OUTCOMES:
Patient engagement in dialogue with clinician about schizophrenia management issues | Measured at visit immediately following intervention/control condition
Clinician satisfaction with interaction with patient | Measured at visit immediately following intervention/control condition
Patient satisfaction with interaction with clinician | Measured at visit immediately following intervention/control condition and at Month 2 post-intervention
Symptoms of psychosis | Measured at Month 2 post-intervention
Symptoms of depression | Measured at Month 2 post-intervention
Quality of life ratings | Measured at Month 2 post-intervention
Adherence to care regimen | Measured at Month 2 post-intervention
Satisfaction with outcomes of care | Measured at Month 2 post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Donald M. Steinwachs, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland